CLINICAL TRIAL: NCT06277388
Title: Hemodynamic Changes and Prognostic Analysis of Patients With Locally Advanced Non-small Cell Lung Cancer During Combined Chemoradiotherapy and Immunotherapy: An Observational Study Based on Dynamic Cardiac Output.
Brief Title: Evaluation of Impedance Cardiography for Assessing Hemodynamic Shifts in Patients With LA-NSCLC During Treatment.
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Clinical Professor, Sun Yat-sen University
Other Study IDs: GASTO-10108
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer; Cardiac Toxicity
Keywords: Non-small Cell Lung Cancer; impedance cardiography; concurrent chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Cardiotoxicity | interventions — Cardiography, Impedance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Impedance cardiography(ICG): The ICG during 6MWT was performed before induction chemo-immunotherapy, before CCRT, and before consolidative immunotherapy for patients with locally advanced NSCLC.
  Interventions: Device: Impedance cardiography

INTERVENTIONS:
Device: Impedance cardiography — The study conducted a 6-minute walk test (6MWT) in a hospital hallway following ATS guidelines. Patients rested for 10 minutes before the test. Impedance measurements were taken before (2 minutes), during (6 minutes), and after (3 minutes) the walk, recording cardio-dynamic parameters with impedance cardiography (ICG).

SUMMARY:
This study aimed to investigate the role of impedance cardiography (ICG) in evaluating hemodynamic changes during the 6-minute walk test (6MWT) in patients with locally advanced non-small cell lung cancer (LA-NSCLC) who underwent combined concurrent chemoradiotherapy (CCRT) and immunotherapy. Additionally, It sought to analyze the predictive significance of cardiac parameters to both treatment toxicity and survival prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. had untreated histologically or cytologically confirmed NSCLC
2. be between the age of 18 and 75
3. had unresectable stage IIIA-IIIC disease, as defined by the AJCC 8th edition staging system
4. had an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0~1
5. had adequate bone marrow function (neutrophil count ≥1.5x109/L, hemoglobin concentration ≥90 g/L, platelet ≥100x109/L), kidney function (serum creatinine clearance ≥50 ml/min) and liver function (serum bilirubin ≤1.5 times upper limit of normal (ULN), aspartate transaminase (AST) and alanine transferase (ALT) ≤2.5 ULN)
6. had a forced expiratory volume in 1 second (FEV1) of ≥0.8L.

Exclusion Criteria:

1. mixed small cell and NSCLC histology
2. life expectancy lower than 12 weeks
3. history of another primary malignancy
4. poorly controlled intercurrent illness
5. female in pregnancy or breast-feeding and any situation not suitable for this study judged by researchers
6. patients with contraindications to 6MWT, including unstable angina pectoris or myocardial infarction within the past month, systolic blood pressure (SBP) over 180mmHg, diastolic blood pressure (DBP) over 100mmHg, muscle strength below grade 3, and severe spasm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced non-small cell lung cancer patients treated by neoadjuvant chemotherapy plus immune checkpoint inhibitors following definitive concurrent chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Estimated)
Dates: Start 2021-06-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Stroke volume（SV） | From enrollment to 2 year after radiotherapy
  The volume of blood ejected from the left ventricle of the heart in one contraction or heartbeat.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang H, Wei J, Zheng Q, Meng L, Xin Y, Yin X, Jiang X. Radiation-induced heart disease: a review of classification, mechanism and prevention. Int J Biol Sci. 2019 Aug 8;15(10):2128-2138. doi: 10.7150/ijbs.35460. eCollection 2019. PMID 31592122
- [Background] Dess RT, Sun Y, Matuszak MM, Sun G, Soni PD, Bazzi L, Murthy VL, Hearn JWD, Kong FM, Kalemkerian GP, Hayman JA, Ten Haken RK, Lawrence TS, Schipper MJ, Jolly S. Cardiac Events After Radiation Therapy: Combined Analysis of Prospective Multicenter Trials for Locally Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2017 May 1;35(13):1395-1402. doi: 10.1200/JCO.2016.71.6142. Epub 2017 Mar 16. PMID 28301264
- [Background] Atkins KM, Rawal B, Chaunzwa TL, Lamba N, Bitterman DS, Williams CL, Kozono DE, Baldini EH, Chen AB, Nguyen PL, D'Amico AV, Nohria A, Hoffmann U, Aerts HJWL, Mak RH. Cardiac Radiation Dose, Cardiac Disease, and Mortality in Patients With Lung Cancer. J Am Coll Cardiol. 2019 Jun 18;73(23):2976-2987. doi: 10.1016/j.jacc.2019.03.500. PMID 31196455
- [Background] Wang K, Eblan MJ, Deal AM, Lipner M, Zagar TM, Wang Y, Mavroidis P, Lee CB, Jensen BC, Rosenman JG, Socinski MA, Stinchcombe TE, Marks LB. Cardiac Toxicity After Radiotherapy for Stage III Non-Small-Cell Lung Cancer: Pooled Analysis of Dose-Escalation Trials Delivering 70 to 90 Gy. J Clin Oncol. 2017 May 1;35(13):1387-1394. doi: 10.1200/JCO.2016.70.0229. Epub 2017 Jan 23. PMID 28113017
- [Background] Lang CC, Agostoni P, Mancini DM. Prognostic significance and measurement of exercise-derived hemodynamic variables in patients with heart failure. J Card Fail. 2007 Oct;13(8):672-9. doi: 10.1016/j.cardfail.2007.05.004. PMID 17923361
- [Background] Lang CC, Karlin P, Haythe J, Lim TK, Mancini DM. Peak cardiac power output, measured noninvasively, is a powerful predictor of outcome in chronic heart failure. Circ Heart Fail. 2009 Jan;2(1):33-8. doi: 10.1161/CIRCHEARTFAILURE.108.798611. PMID 19808313
- [Background] Janssen-Heijnen ML, Schipper RM, Razenberg PP, Crommelin MA, Coebergh JW. Prevalence of co-morbidity in lung cancer patients and its relationship with treatment: a population-based study. Lung Cancer. 1998 Aug;21(2):105-13. doi: 10.1016/s0169-5002(98)00039-7. PMID 9829544